CLINICAL TRIAL: NCT03899831
Title: A Randomized Clinical Trial of a Structured Function-Based Elopement Treatment Program
Brief Title: Structured Function-Based Elopement Treatment Program
Acronym: FBET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Autism Speaks (Other)
Responsible Party: Principal Investigator, Mindy Scheithauer, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00108995
Record Dates: First submitted 2019-04-01; First posted 2019-04-02 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Autism Spectrum Disorder
Keywords: Elopement
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to FBET or PEP in a 1:1 ratio using random permuted blocks of size 2 and 4. After Wk 16, participants in the PEP group will be offered the FBET.
Who Masked: Outcomes Assessor
Masking Description: Outcome measures will be administered by a blinded independent evaluator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Function-Based Elopement Treatment (FBET) (Experimental): Participants in this group will receive Function-Based Elopement Treatment (FBET) for 16 weeks.
  Interventions: Behavioral: Function-Based Elopement Treatment (FBET)
- Parent Education Program (PEP) (Active Comparator): Participants in this group will take part in a parent education program (PEP) for 16 weeks.
  Interventions: Behavioral: Parent Education Program (PEP)

INTERVENTIONS:
Behavioral: Function-Based Elopement Treatment (FBET) — The Function-Based Elopement Treatment (FBET) includes 12 appointments over 16 weeks. FBET focuses on parent-training, with the parent implementing procedures with therapist support. The goals of FBET are:
  * to create a safer environment
  * teach adaptive skills to replace elopement
  * arrange the environment and rewards to reduce elopement
  * and teach caregivers how to respond if elopement occurs Psychoeducation is emphasized, including discussions of elopement as a learned behavior, reinforcement, functions of elopement, extinction, and descriptions of treatment components. The FBET manual includes scripted text, examples, caregiver completed activities, and checks for understanding.
  Arms: Function-Based Elopement Treatment (FBET)
Behavioral: Parent Education Program (PEP) — The Parent Education Program (PEP) will include 12 appointments over 16 weeks, focused on general education about autism spectrum disorder and resources about elopement prevention. PEP will be administered by a Board Certified Behavior Analyst (BCBA). Participants randomized to the PEP study arm can receive the FBET intervention after completing the 16 week study period.
  Arms: Parent Education Program (PEP)

SUMMARY:
This study aims to extend the researchers' prior work on Function-Based Elopement Treatment (FBET) with a randomized controlled trial to evaluate the efficacy of FBET in 76 children with autism spectrum disorder (ASD) and elopement. Participants will be randomized to FBET or an active control group receiving a parent education program (PEP). Each study arm will include 12 appointments over 16 weeks and will be administered by a Board Certified Behavior Analyst (BCBA).

DETAILED DESCRIPTION:
Elopement (running/wandering away from supervision) affects nearly 50% of children with ASD and is a contributor to the fact that children with ASD have nearly double the premature death rate of their typically developing peers. Existing interventions, such as prevention kits, increase safety by decreasing elopement opportunities (e.g., locking doors), but do not necessarily decrease attempts. Given that a single successful attempt can be fatal, the fact that prevention-only strategies cannot eliminate elopement means that other treatment approaches are necessary. Interventions based in applied behavior analysis (ABA) have been successful in reducing elopement attempts. ABA relies on function-based treatments, which start with assessment to identify why an individual elopes (i.e., its function). Common functions of elopement include accessing attention (e.g., parent's reaction), preferred items (e.g., toys), or escape from nonpreferred situations (e.g., leaving a store). Function is crucial, as common strategies may be contraindicated based on function. For example, a caregiver may pick up a child and discuss safety after elopement. Unfortunately, this may reinforce elopement, and make it worse, if the function for that child is to gain attention. Key elements of function-based treatments include preventing delivery of the functional reinforcer following elopement (i.e., extinction) and teaching an appropriate means of accessing it instead.

While there is support in the literature for function-based treatments, it has relied on small sample sizes. In the largest elopement treatment study to date, the researchers demonstrated significant improvements based on clinical outcomes. However, even this study was relatively small (N=11) and lacked a control group. The bulk of research supporting these interventions has also been conducted in specialized treatment centers by doctoral level professionals. This is in contrast to the majority of ABA services delivered by Master level Board Certified Behavior Analysts (BCBAs) operating in community settings. Thus, even if ABA-based interventions are efficacious, their generality and community viability remain unknown. Finally, research has evaluated either prevention strategies or function-based interventions, while studies combining these are strikingly absent.

A randomized controlled trial designed to test the efficacy of a structured, exportable intervention for elopement with prevention strategies and function-based interventions has not been conducted, but is critical for several reasons. First, rigorous studies with a control group and sufficient sample size are needed for function-based treatments to be widely accepted as empirically supported. Second, evaluation of a manualized intervention combining these approaches implemented in a community context will demonstrate the viability outside of specialized clinics. A manualized treatment can serve as a much needed resource for community providers faced with treating elopement. The researchers have developed a manualized, parent-mediated intervention called Function-Based Elopement Treatment (FBET). In a pilot feasibility study the researchers evaluated FBET with 24 children with ASD (age 4 to 12), who were randomly assigned to FBET (n=12) or a waitlist (n=12).

In this study, participants will be randomized to receive the FBET intervention or PEP for 16 weeks. Participants in the PEP study arm will be offered the opportunity to have the FBET intervention at the end of the 16 week study period. The study aims are to:

Aim 1: Evaluate whether FBET is superior to PEP in reducing elopement in 76 children (age ≥ 4 to ≤ 12) with ASD after 16 weeks of treatment using the Aberrant Behavior Checklist-Hyperactivity subscale (ABC-H).

Aim 2: Evaluate two key secondary outcomes (at Wk 16): a) the independent evaluator ratings on the Clinical Global Impression-Improvement rating (CGI-I) and b) home safety, based on the percentage of prevention items endorsed on the home elopement safety checklist (HESC).

Aim 3: Evaluate whether direct observation of elopement, based on parent data on elopement frequency for one week leading up to each assessment point, demonstrates a significant decrease in the FBET compared to PEP participants.

Aim 4: Evaluate whether gains made in the FBET group are maintained after treatment (at Wk 28, using the ABC-H, HESC, and CGI-I)

Exploratory Aim 1: To evaluate the impact of FBET on disruptive behavior using the ABC-Irritability subscale

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 4 to ≤ 12
* diagnosis of ASD, confirmed by clinical characterization of an Autism Diagnostic Observation Schedule (ADOS), Autism Diagnostic Interview-Revised (ADI-R), or Childhood Autism Rating Scale-Second Edition (CARS-2), cognitive (e.g., Differential Abilities Scale [DAS], Mullen Scales of Early Learning [MSEL or Mullen]), and adaptive assessments (Vineland Adaptive Behavior Scales-Third Edition [Vineland-3])
* chief complaint of elopement
* an ABC-H score > 18

Exclusion Criteria:

* caregivers who report they cannot reliably attend appointments
* ongoing or planned treatment that would likely impact elopement
* challenging behavior that should be treated prior to elopement

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Change in Aberrant Behavior Checklist - Hyperactivity (ABC-H) Subscale Score | Baseline, Week 16
  Elopement will be measured by the hyperactivity subscale of the Aberrant Behavior Checklist (ABC-H). The full ABC is a 58-item caregiver completed measure with 5 subscales. It is used extensively with children with ASD in clinical trials and has demonstrated validity and reliability with this population. Although the ABC-H targets hyperactivity, there are several items directly related to elopement. The hyperactivity subscale includes 16 items that are answered on a scale of 0 (not a problem) to 3 (severe problem). Scores for this subscale range from 0 to 48, where higher scores indicate a higher severity of hyperactivity.

SECONDARY OUTCOMES:
Change in Clinical Global Impression - Improvement (CGI-I) Score | Week 16
  CGI-I asks an independent evaluator to rate the degree of improvement, compared to the last visit, on a scale of 1 (very much improved) through 4 (no change) to 7 (very much worse).
Change in Home Elopement Safety Checklist (HESC) Score | Baseline, Week 16
  The Home Elopement Safety Checklist (HESC) is a 22-item instrument listing steps to prevent elopement (e.g., locks, alarms) and decrease safety risk if elopement were to occur (e.g., purchasing identification bracelets). Parents indicate if each item has been completed or not and the percentage of completed items is the total safety score. The a higher percentage means that more safety elements have been implemented in order to reduce elopement or to increase the child's safety if they do elope.
Direct observation of elopement frequency | Baseline, Week 16
  The frequency of elopement will be assessed based on parent data on elopement frequency for one week leading up to each assessment point.
Change in Aberrant Behavior Checklist - Hyperactivity (ABC-H) Subscale Score | Week 16, Week 28
  To evaluate whether gains made in the FBET group are maintained after treatment, the ABC-H will be repeated at the Week 28 follow up visit. Elopement will be measured by the hyperactivity subscale of the Aberrant Behavior Checklist (ABC-H). The full ABC is a 58-item caregiver completed measure with 5 subscales. It is used extensively with children with ASD in clinical trials and has demonstrated validity and reliability with this population. Although the ABC-H targets hyperactivity, there are several items directly related to elopement. The hyperactivity subscale includes 16 items that are answered on a scale of 0 (not a problem) to 3 (severe problem). Scores for this subscale range from 0 to 48, where higher scores indicate a higher severity of hyperactivity.
Change in Clinical Global Impression - Improvement (CGI-I) Score | Week 28
  To evaluate whether gains made in the FBET group are maintained after treatment, the CGI-I will be repeated at the Week 28 follow up visit. CGI-I asks an independent evaluator to rate the degree of improvement, compared to the last visit, on a scale of 1 (very much improved) through 4 (no change) to 7 (very much worse).
Change in Home Elopement Safety Checklist (HESC) Score | Week 16, Week 28
  To evaluate whether gains made in the FBET group are maintained after treatment, the HESC will be repeated at the Week 28 follow up visit. The HESC is a 22-item instrument listing steps to prevent elopement (e.g., locks, alarms) and decrease safety risk if elopement were to occur (e.g., purchasing identification bracelets). Parents indicate if each item has been completed or not and the percentage of completed items is the total safety score. The a higher percentage means that more safety elements have been implemented in order to reduce elopement or to increase the child's safety if they do elope.

OTHER OUTCOMES:
Change in Aberrant Behavior Checklist - Irritability (ABC-I) Scale Score | Baseline, Week 16
  This exploratory aim evaluates the impact of FBET on disruptive behavior, as measured by the irritability subscale of the Aberrant Behavior Checklist (ABC-I). The full ABC is a 58-item caregiver completed measure with 5 subscales. The irritability subscale includes 15 items that are answered on a scale of 0 (not a problem) to 3 (severe problem). Scores for this subscale range from 0 to 45, where higher scores indicate increased severity of disruptive behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Mindy Scheithauer, PhD, Principal Investigator — Emory University
Locations (1):
- Marcus Autism Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) collected during the trial, will be available for sharing following deidentification.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: IPD will be shared beginning 3 months after article publication and ending 5 years following publication.
Access Criteria: IPD will be shared with researchers providing a methodologically sound proposal in order to achieve the aims in the proposal or for meta-analyses. Proposals should be directed to Mindy.Scheithauer@choa.org. To gain access, data requestors may need to sign a data access agreement. Proposals may be submitted up to 5 years following article publications.